CLINICAL TRIAL: NCT03799016
Title: An Observational Study on Incidence, Natural History and Treatment Patterns of Venous Thromboembolism in Taiwan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18787
Record Dates: First submitted 2018-10-25; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The research question addressed by this study is primarily on the clinical epidemiology of VTE in Taiwan. The study aims to estimate the incidence of VTE and describe natural history of VTE, including long term clinical outcomes in adult Taiwanese population, utilizing population-based electronic health data in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* The source population was the adult population in Taiwan. The legal age for definition as an adult (without additional research ethics review requirement) in Taiwan is 20; therefore all National Health Insurance (NHI) enrollees age 20 or older at any time during the study period were evaluated for VTE.

Exclusion Criteria:

* Person-time before an eligible subject turned 20 were not evaluated.
* Study subjects having inconsistent data on gender and unrealistic date of birth (birth year before 1890 and after 2015) were identified and excluded from the analysis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 104215 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Incident VTE | 4 years
  Incident VTE cases were those who had a first VTE diagnosis after 1 January 2005 and with at least 5 years of look-back period. Those with a first VTE diagnosis less than 5 years of look-period were considered as undetermined VTE cases.
Potential risk factors that occurred before the incident VTE events | 4 years
  Events during the 3 months before the first VTE recurrence will be described. Potential risk factors that will be evaluated include age, gender, and treatment regimen for VTE, adherence to treatment regimen, concomitant medications, and comorbidity. The analysis will be stratified by the nature of the first VTE (provoked and unprovoked). Due to the unknown number of repeated recurrence and complex clinical nature of patients with multiple VTE recurrence, risk factors for multiple recurrences will be evaluated at a less detailed level than that for the first recurrence.
Usage patterns of anticoagulants among incident VTE patients were evaluated during incident VTE hospital admission and after discharge | 4 years
All-cause mortality | 4 years
  All deaths before 31 December 2014 among the incident VTE patients were identified through the mortality records. Patients were followed from incident VTE index date, and the patients were censored on 31 December 2014 or termination of NHI coverage without further medical or mortality records. If the patient died during the same hospitalization during the incident VTE, the death date was defined as the discharge date of that specific hospitalization.
Major bleeding | 4 years
  Major bleeding (intracranial bleed and gastrointestinal bleed) was the major morbidity of interest and incident VTE patients were followed from incident VTE index date till 31 December 2014, death or termination of NHI coverage without any further medical records. Patients died during the incident VTE hospitalization were excluded for major bleeding follow up.
Recurrent VTE | 4 years
  Recurrent VTE events after the incident VTE diagnosis were evaluated during the follow-up period through 31 December 2014 or until the patient died or NHI coverage terminated without any further medical records after the termination. The same VTE operational definitions according to different algorithm in incident VTE were consistently applied in recurrent VTE.
Adherence of oral anticoagulant treatment was also evaluated with the calculation of MPR within 6 months and 12 months after discharge. | Up to 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Taipei, Taiwan